CLINICAL TRIAL: NCT03966924
Title: The PREFORM Study: An Exploratory, Single-Center Study to Evaluate the Safety and Efficacy of Rotational Fractional Resection on Submental Contouring and Optimal Peri-Procedure Regimen for Accelerated Recovery
Brief Title: The PREFORM Study: Rotational Fractional Resection for Submental Contouring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recros Medica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-0007
Record Dates: First submitted 2019-03-19; First posted 2019-05-29 (Actual); Results first posted 2021-02-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2020-01

CONDITIONS: Skin Laxity; Lipodystrophy
Keywords: submental; laxity; lipodystrophy
MeSH Terms: conditions — Cutis Laxa; Lipodystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Rotational fractional resection (1.5mm Diameter Device) (Experimental): Single treatment of skin resection and with and without focal lipectomy (removal of loose skin and fat)
  Interventions: Device: Rotational fractional resection (1.5mm Diameter Device)

INTERVENTIONS:
Device: Rotational fractional resection (1.5mm Diameter Device) — Single treatment of skin resection and with and without focal lipectomy (removal of loose skin and fat)

SUMMARY:
This study will evaluate the safety and efficacy of rotational fractional resection (RFR) to improve neck contouring. Rotational fractional resection is used to remove loose skin and fat.

DETAILED DESCRIPTION:
This is a prospective, single-center, single-arm (non-randomized), interventional cohort, non-significant risk (NSR) study designed to investigate the efficacy and safety of Rotational Fractional Resection (skin resection and focal lipectomy) in patients with moderate to severe submental skin laxity. The total duration of study participation for each subject is approximately up to 4 months for each subject from the screening visit to the exit visit. The follow-up period will be approximately 3 months after the procedure. Eligible subjects will complete a total of 11 study visits: screening, procedure, and follow-up visits at 1, 4, 7, 14, 21, 30, 45, 60, and 90 days post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* At least 30 years old
* Moderate to severe submental laxity
* Up to moderate submental lipodystrophy
* Agree to maintain weight (±5%) for the duration of the study

Exclusion Criteria:

* Previous intervention to treat submental fat or skin laxity
* Use of aspirin, ibuprofen, naproxen, or Vitamin E within 14 days of the procedure
* Severe acne, cystic acne or acne scars on neck
* Trauma of chin or neck area
* Skin infection or rash on neck
* Psoriasis, hyperpigmentation, eczema, rosacea or vitiligo
* History of scarring
* Body mass index (BMI) >30
* Clinically significant bleeding disorder
* Anemia, kidney disease, or liver disease

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin McIntosh, Study Director — Recros Medica
Locations (1):
- Steve Yoelin, MD Medical Associates, Inc., Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rotational Fractional Resection (1.5mm Diameter Device)
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rotational Fractional Resection (1.5mm Diameter Device)
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 57 [55 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Submental Skin Laxity Scale score [Count of Participants; unit: Participants] — Measurement of submental skin laxity on a 5 point scale: grades 0-4. Subjects were enrolled with moderate or severe submental skin laxity.
  Participants
    Moderate | 1
    Severe | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had at Least One Grade Improvement on the Submental Skin Laxity Scale
Description: Physician investigator rated the submental laxity using the Submental Skin Laxity scale (0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe)
Time Frame: 90 days post treatment
Population: Number of participants with at least a one grade improvement on the Submental Skin Laxity Scale
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Fractional Resection (1.5mm Diameter Device)
Number analyzed (Participants) | 2
Participants | 2

2. Secondary Outcome: Number of Participants Who Were Satisfied With the Appearance of Their Neck and Jawline
Description: Subjects rated their satisfaction of the appearance of their neck and jawline on a Subject Satisfaction Questionnaire. Results reflect subjects who were satisfied ("somewhat satisfied," "satisfied," or "very satisfied").
Time Frame: 90 days post treatment
Population: Number of Participants Who Were Satisfied With the Appearance of Their Neck and Jawline
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Fractional Resection (1.5mm Diameter Device)
Number analyzed (Participants) | 2
Participants | 2

3. Secondary Outcome: Number of Participants With a One Grade Improvement on the Submental Lipodystrophy Scale
Description: Comparison of the submental fat before and after procedure using the Submental Skin Lipodystrophy scale (0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe)
Time Frame: 90 days post treatment
Population: 1 grade improvement (Mild to None)
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Fractional Resection (1.5mm Diameter Device)
Number analyzed (Participants) | 2
Participants | 2

ADVERSE EVENTS:
Time Frame: 90 days post treatment
Arm/Group | Rotational Fractional Resection (1.5mm Diameter Device)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotational Fractional Resection (1.5mm Diameter Device) (N=2)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) — Skin irritation near procedure area as a result of a silicone pad

LIMITATIONS AND CAVEATS:
This study evaluated 1.5mm diameter skin resections, the first-generation prototype, in the submental area.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/24/NCT03966924/Prot_000.pdf